CLINICAL TRIAL: NCT01318863
Title: A Normal Donor Sample Collection Study in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AST-015
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Normal Volunteers
Keywords: aged matched normal control samples

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
More than one site will participate in the collection of blood and urine samples from healthy adult subjects. These samples will be used for future testing to serve as aged-matched normal controls and to establish normal reference ranges in the development of new invitro diagnostic devices.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults (age ≥ 21 years)
* Provide written informed consent for study participation

Exclusion Criteria:

* Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days;
* Any known or suspected significant chronic medical conditions (such as diabetes, coronary artery disease, renal insufficiency, hypertension, hypercholesterolemia, chronic inflammatory diseases [e.g., rheumatoid arthritis], cancer, etc);
* Trauma-related surgery within the last 6 months;
* Any surgery, hospitalization or institutionalization (such as in a nursing home) during the previous 3 months;
* Received any blood product transfusion within the previous 2 months;
* Pregnant women or children;
* Prisoners or institutionalized individuals;
* Already provided blood or urine samples for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Apex Research Institute, Santa Ana, California
  - Clinical Research Consortium, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Gray, Tennessee
  - Memphis, Tennessee
  - Research Across America, Dallas, Texas